CLINICAL TRIAL: NCT02308618
Title: Achilles Tendon Rupture: Comparative Study Between Two Rehabilitation Programs.
Brief Title: Rehabilitation Programs After Achilles Tendon Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFRGS - 2007882
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Rupture of Achilles Tendon; Immobility Response, Tonic; Rupture, Spontaneous
Keywords: Achilles tendon rupture; Rehabilitation; Immobilization; Muscle architecture; Functionality; Neuromuscular parameters; Weight-Bearing
MeSH Terms: conditions — Immobility Response, Tonic; Rupture, Spontaneous | interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Traditional Immobilization (Experimental): 45 days of plaster cast immobilization After the immobilization period, subjects received instructions on how to perform a home-based exercise program
  Interventions: Other: Traditional Immobilization
- Early mobilization (Experimental): Six weeks of physical therapy program
  Interventions: Other: Early Mobilization
- Control (No Intervention): Subjects had no history of lower limb injury, and were matched in age and anthropometric measurements to subjects that performed physical rehabilitation and to subjects that remained immobilized.

INTERVENTIONS:
Other: Traditional Immobilization — After surgery subjects were immobilized in a plaster cast, with the ankle positioned in gravitational equinus; weight bearing was not allowed. Two weeks post-operatively, the cast was removed and the patient was immobilized with a new plaster cast, with the ankle in the same position. Four weeks post-operatively, the ankle was plastered in neutral position (i.e. with the sole of the foot perpendicular to the shank), and weight bearing was encouraged. Six weeks post-operatively, the plaster cast was removed
  The home exercise program consisted of active exercises and stretches to improve ankle range of motion, and resistance and balance exercises
  Other Names: Plaster cast immobilization
  Arms: Traditional Immobilization
Other: Early Mobilization — The physical therapy started two weeks after the surgery and lasted six weeks, during which a removable brace was used. Therapy sessions, three times per week in the six-week period, included one to two hours of exercises for regaining range of motion and muscular endurance.
  Other Names: Accelerated rehabilitation
  Arms: Early mobilization

SUMMARY:
The purpose of this study is to evaluate the effects of early mobilization versus traditional immobilization rehabilitation programs after surgical Achilles tendon repair on the mechanical (torque-angle and torque-velocity relationships) and electrical (neuromuscular activation) properties of the plantar- and dorsiflexor muscles, gastrocnemius medialis morphology (muscle architecture), functional performance, and the mechanical and material properties (force-elongation and stress-strain relationships) of the injured and uninjured Achilles tendon.

The hypothesis is that the early mobilization could reduce the deleterious effects of the joint immobilization and improve the tendon healing.

DETAILED DESCRIPTION:
Participants were allocated into one of two intervention groups (traditional immobilization or early mobilization).

Traditional immobilization group (45 days of plaster cast immobilization; after the immobilization period, subjects received instructions on how to perform a home-based exercise program)

Early mobilization (six weeks of physical therapy program; three times per week; one to two hours of exercises for regaining range of motion and muscular endurance)

Control group (subjects had no history of lower limb injury, and were matched in age and anthropometric measurements to subjects that performed physical rehabilitation and to subjects that remained immobilized.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Achilles tendon rupture

Exclusion Criteria:

* arterial insufficiency
* diabetes
* autoimmune disease
* patients who used systemic antibiotics or steroids or showed any other clinical contraindication to perform maximum voluntary contractions on a dynamometer.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Torque change | Torque was measured 3 times during the study: three, six and more than 12 months after surgical repair.
  Torque is an expression of the muscular strength and was assessed by dynamometry

SECONDARY OUTCOMES:
Ankle range of motion change | Ankle range of motion was measured 5 times during the study: 15 days, 45 days, three, six and more than 12 months after surgical repair.
  Ankle range of motion was assessed by goniometry during active and passive dorsiflexion and plantar flexion.
Muscular architecture change | Muscle architecture was measured 4 times during the study: 45 days, three, six and more than 12 months after surgical repair.
  Muscular architecture (muscle thickness, pennation angle and fascicle length) was assessed by ultrasonography
Plantarflexor muscle volume change | Plantarflexor muscle volume was assessed 4 times during the study: 45 days, three, six and more than 12 months after surgical repair.
  Plantarflexor muscle volume was estimated from calf muscle thickness and limb length using the equation proposed by Miyatani et al. 2004.

OTHER OUTCOMES:
Muscular electrical activation change | Muscular electrical activation was measured 3 times during the study: three, six and more than 12 months after surgical repair
  Electrical activation was assessed by electromyography (EMG)
Tendon mechanical and material properties change | Tendon mechanical and material properties were measured 3 times during the study: three, six and more than 12 months after surgical repair.
  Tendon mechanical and material properties were assessed by Achilles tendon elongation (measured by ultrasound) during isometric plantar flexion ramp contraction as a function of ankle joint torque.
Functional performance change | Functional performace was measured 3 times during the study: three, six and more than 12 months after surgical repair
  Functional performance was assessed by functional tests (standing heel-rise, time up and go and jump tests) and AOFAS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil